CLINICAL TRIAL: NCT04026178
Title: A 36-Month, Multicenter, Open Label Phase 4 Study to Evaluate the Immunogenicity of Daily SC Metreleptin Treatment in Patients With Generalized Lipodystrophy
Brief Title: Immunogenicity of Metreleptin in Patients With Generalized Lipodystrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEGR-734-401
Record Dates: First submitted 2018-10-30; First posted 2019-07-19 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Generalized Lipodystrophy
Keywords: Immunogenicity; Antibodies; Lipodystrophy
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized; Lipodystrophy | interventions — metreleptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metreleptin (Experimental): Subjects will receive prescribed dosage of metreleptin as indicated in the USPI Patients (males and females) ≤ 40 kg: 0.06mg/kg Male patients > 40 kg: 2.5mg Female patients > 40 kg: 5mg
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — Subjects will receive prescribed dosage of metreleptin as indicated in the USPI

SUMMARY:
MYALEPT™ (metreleptin) has been approved as an adjunct to diet as replacement therapy to treat the complications of leptin deficiency in patients with congenital or acquired generalized lipodystrophy (MYALEPT Prescribing Information). This study is a multicenter, open-label, Phase 4 trial to provide an assessment of the immunogenicity associated with metreleptin and of any major potential risks due to development of antibodies to metreleptin. The study is being conducted to comply with a postmarketing requirement.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures. If <18 years of age, has a parent or guardian able to read, understand, and sign the Informed Consent Form (ICF) and a Child Assent form, communicate with the Investigator, and understand and comply with protocol requirements. Adolescent patients must also read and understand the Child Assent Form. If the child is too young or unable to read, then the Child Assent form must be explained to the child.
2. Female and/or male patients ≥1 years of age.
3. Physician-confirmed diagnosis of congenital or acquired generalized lipodystrophy and will begin treatment with MYALEPT for the first time.
4. Negative pregnancy test (urine or serum) for female patients of childbearing potential.
5. Female patients of childbearing potential must be 1 year postmenopausal, surgically sterile, or be willing to use an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent). In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.
6. Male patients must be surgically sterile or be willing to use an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent).
7. Patients who are blood donors should not donate blood during the study and for 3 months following their last dose of metreleptin.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Aegerion staff and/or staff at the study site.)
2. Previous treatment with metreleptin.
3. Participation in another clinical study with an investigational product during the last 6 months.
4. Patients with prior severe hypersensitivity reactions to metreleptin or to any of the product components.
5. Known to have tested positive for human immunodeficiency virus, are immunocompromised, or are receiving immunomodulatory drugs.
6. Known history of drug or alcohol abuse within 1 year of screening.
7. Creatinine clearance <30 mL/min using institutional standards:

   e.g., calculated using Cockcroft-Gault formula for patients ≥18 years of age; calculated using Schwartz equation for patients <18 years of age.
8. For women only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
9. Any condition where, in the opinion of the Investigator, participation in this study may pose a significant risk to the patient or could render the patient unable to successfully complete the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Boylan, Study Director — Aegerion Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - Univ. Alabama-Birmingham, Birmingham, Alabama
  - Ochsner Clinic, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Endocrinology Research Associates, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University Texas Southwestern INT, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
only IPD that underly results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: A copy of data generated at the study site will be provided to individual sites after the overall publication by the sponsor is completed and submitted

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 4 centers in the US. Prescribing Investigators for this study were those who were certified under REMS for MYALEPT prescription and able to ensure prescription of metreleptin was as per the USPI.
Pre-assignment Details: At Screening, consenting patients were assessed to ensure that they met eligibility criteria. The informed consent and health insurance portability and accountability act Authorization forms were signed prior to performing any Protocol-required procedures. The assessments conducted at the Screening Visit. When all Screening results were available, individuals were notified of their eligibility status.
Groups:
- Metreleptin: Subjects will receive prescribed dosage of metreleptin as indicated in the USPI:
  Patients (males and females) ≤ 40 kg: 0.06mg/kg Male patients > 40 kg: 2.5mg Female patients > 40 kg: 5mg
Period: Overall Study
Arm/Group | Metreleptin
Started | 11
Completed | 7
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Metreleptin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Lipodystrophy diagnosis [Count of Participants; unit: Participants] — Population: 11 GL: 6 Congenital Generalized Lipodystrophy, and 5 Acquired Generalized Lipodystrophy
  Participants
    Congenital Generalised Lipodystrophy | 6
    Acquired Generalised Lipodystrophy | 5
Medical History [Count of Participants; unit: Participants]
  Hypertriglyceridemia | 8
  Diabetes | 7
  Pancreatitis | 5
  Hypertension | 4
  Hepatic steatosis | 3
  Polycystic ovary syndrome | 2
  Proteinuric | 2
  Hepatic cirrhosis | 1

OUTCOME MEASURES:

1. Secondary Outcome: Assess 2 Methods of Measuring in Vitro NAb Activity to Metreleptin.
Description: The percent (standard error) of patients with a positive result was compared for the RB NAb assay and the cell-based NAb assay over time.
Time Frame: 36 months
Population: Only ADA+ participants were analysed for neutralizing activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Metreleptin
Number analyzed (Participants) | 10
Participants
  NAb cell based+ | 1
  NAb receptor blocking+ | 10

2. Secondary Outcome: Evaluate the Safety and Tolerability in Relation to the Development of or Absence of Anti-metreleptin and Anti-HuL Binding ADAs, and/or in Vitro NAb Activity to Metreleptin in Patients With CGL or AGL
Description: Serious adverse events (SAEs), AEs leading to discontinuation, loss of response (as assessed by glycated hemoglobin (HbA1c) and serum triglycerides), severe infections and/or sepsis, standard laboratory tests, and vital signs over time.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metreleptin
Number analyzed (Participants) | 11
Participants
  All AE: AEs leading to discomntinuation | 11
  SAE: AEs leading to discomntinuation | 7
  AEs leading to discontinuation: AEs leading to discomntinuation | 1
  Severe infections and/or sepsis: AEs leading to discomntinuation | 2
  Blood Triglycerides increased: AEs leading to discomntinuation | 3
  Glycosylated haemoglobin increased: AEs leading to discomntinuation | 1

3. Other Pre Specified Outcome: Evaluate the Efficacy With Daily Metreleptin in Patients With GL
Description: Change from Baseline in HbA1c over time.
Time Frame: 36 months
Population: Only subjects who reached the visits (Month 12, 24 ,36) were included in the analysis
Measure: Median (Full Range); unit: Percentage
Arm/Group | Metreleptin
Number analyzed (Participants) | 11
Percentage
  Absolute change in HbA1c from baseline to Month 12: number analyzed (Participants) | 8
  Absolute change in HbA1c from baseline to Month 12 | -0.3 [-6.5 to 2.3]
  Absolute change in HbA1c from baseline to Month 24: number analyzed (Participants) | 8
  Absolute change in HbA1c from baseline to Month 24 | -0.5 [-7.2 to 1.8]
  Absolute change in HbA1c from baseline to Month 36: number analyzed (Participants) | 7
  Absolute change in HbA1c from baseline to Month 36 | -0.7 [-7.3 to 1.9]

4. Primary Outcome: Evaluate the Immunogenicity Associated With Daily Subcutaneous (SC) Metreleptin Treatment in Patients With Congenital Generalized Lipodystrophy (CGL) or Acquired Generalized Lipodystrophy (AGL).
Description: Anti-metreleptin, anti-human leptin (HuL) binding antidrug antibody (ADA) titers over time. Category of in vitro cell-based neutralizing antibody (NAb) activity to metreleptin, and titer in the receptor blocking (RB) NAb assay in ADA positive samples over time.
Time Frame: 36 months
Population: Only ADA positive participants were analysed for neutralizing activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Metreleptin
Number analyzed (Participants) | 11
Participants
  ADA positive: ADA+ | 10
  NAb cell based +: number analyzed (Participants) | 10
  NAb cell based +: ADA+ | 1
  NAb receptor blocking+: number analyzed (Participants) | 10
  NAb receptor blocking+: ADA+ | 10

5. Other Pre Specified Outcome: Evaluate the Efficacy With Daily Metreleptin in Patients With GL
Description: Percent change from Baseline in fasting triglycerides over time.
Time Frame: 36 months
Population: Only subjects who reached the visits (Month 12, 24 ,36) were included in the analysis
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Metreleptin
Number analyzed (Participants) | 11
Percent Change
  Precent change in triglycerides from baseline to Month 12: number analyzed (Participants) | 9
  Precent change in triglycerides from baseline to Month 12 | -49.68 [-91.26 to 174.77]
  Precent change in triglycerides from baseline to Month 24: number analyzed (Participants) | 8
  Precent change in triglycerides from baseline to Month 24 | -46.72 [-92.25 to 593.01]
  Precent change in triglycerides from baseline to Month 36: number analyzed (Participants) | 7
  Precent change in triglycerides from baseline to Month 36 | -58.12 [-98.55 to -22.16]

ADVERSE EVENTS:
Time Frame: From signing the ICF up until either the last scheduled Follow-up Visit (36 months) or at least 4 weeks after the last dose of study medication in the case of an early termination
Arm/Group | Metreleptin
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metreleptin (N=11)
COVID-19 (Infections and infestations) | 1 — COVID-19 infection, not related to metreleptin
Autoimmune hepatitis (Hepatobiliary disorders) | 1 — Exacerbation of autoimmune hepatitis, not related to metreleptin
Pancreatitis relapsing (Gastrointestinal disorders) | 1 — Recurrent pancreatitis, not related to metreleptin
Osteomyelitis (Infections and infestations) | 1 — Osteomyelitis (fifth digit of left hand), not related to metreleptin
Sepsis (Infections and infestations) | 1 — Sepsis, not related to metreleptin
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 — Miscarriage, not related to metreleptin
Constipation (Gastrointestinal disorders) | 1 — Constipation, not related to metreleptin
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metreleptin (N=11)
Anemia (Blood and lymphatic system disorders) | 1 — Anemia, not related to metreleptin
Cardiac failure (Cardiac disorders) | 1 — Heart failure, not related to metreleptin
Cerumen impaction (Ear and labyrinth disorders) | 1 — Bilateral impacted cerumen, not related to metreleptin
Cataract (Eye disorders) | 1 — Bilateral cataracts, not related to metreleptin
Abdominal pain (Gastrointestinal disorders) | 3 — Abdominal pain, not related to metreleptin
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhea (General disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 — Chronic pancreatitis, not related to metreleptin
Vomiting (Gastrointestinal disorders) | 1 — Vomiting, not related to metreleptin
Injection site haemorrhage (General disorders) | 1 — Very small blead of blood after one injection, not related to metreleptin
Peripheral swelling (General disorders) | 1 — Left leg swelling, not related to metreleptin
Ocular icterus (Hepatobiliary disorders) | 1 — Jaundice eyes, not related to metreleptin
Bacterial vaginosis (Infections and infestations) | 1 — Bacterial vaginosis, not related to metreleptin
Chlamydial infection (Infections and infestations) | 1 — Chlamydia, not related to metreleptin
COVID-19 (Infections and infestations) | 4 — COVID-19, not related to metreleptin
Croup infectious (Infections and infestations) | 1 — Croup, not related to metreleptin
Infectious mononucleosis (Infections and infestations) | 1 — Mononucleosis, not related to metreleptin
Influenza (Infections and infestations) | 1 — Flu, not related to metreleptin
Respiratory syncytial virus infection (Infections and infestations) | 1 — RSV infection, not related to metreleptin
Sinusitis (Infections and infestations) | 1 — Sinus infection, not related to metreleptin
Tonsilitis (Infections and infestations) | 1 — Tonsilitis, not related to metreleptin
Urinary tract infection (Infections and infestations) | 1 — Urinary tract infection, not related to metreleptin
Viral infection (Infections and infestations) | 1 — Viral illness, not related to metreleptin
Fall (Injury, poisoning and procedural complications) | 1 — Fall, not related to metreleptin
Foot fracture (Injury, poisoning and procedural complications) | 1 — Foot fracture, not related to metreleptin
Hand fracture (Injury, poisoning and procedural complications) | 1 — LEFT HAND FRACTURES IN 3 PLACES - HAND HIT WALL IN INDOOR SOCCER GAME, not related to metreleptin
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 2 — Pregnancy
Skin laceration (Injury, poisoning and procedural complications) | 1 — STITCHES IN CHIN FOR LACERATION, not related to metreleptin
Blood bilirubin increased (Investigations) | 1 — Elevated bilirubin level, not related to metreleptin
Blood cholesterol increased (Investigations) | 1 — High cholesterol, not related to metreleptin
Blood pressure increased (Investigations) | 1 — Elevated blood pressure, not related to metreleptin
Blood triglycerides increased (Investigations) | 2 — Elevated triglyceride level, not related to metreleptin
Glycosylated haemoglobin increased (Investigations) | 1 — High HbA1c, not related to metreleptin
Liver function test increased (Investigations) | 1 — Increased liver function tests, not related to metreleptin
Hyperglycemia (Metabolism and nutrition disorders) | 1 — Hyperglycemia, not related to metreleptin
Hyperkalemia (Metabolism and nutrition disorders) | 1 — Hyperkalemia, not related to metreleptin
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 — Left shoulder pain, not related to metreleptin
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — BASAL CELL CARCINOMA, MULTIPLE (RIGHT SHOULDER, RIGHT UPPER ARM, RIGHT LOWER BACK) NO SIZE PROVIDED, not related to metreleptin
Hypoesthesia (Nervous system disorders) | 1 — Increasing in leg numbness, not related to metreleptin
Motor dysfunction (Nervous system disorders) | 1 — Worsening motor dysfunction, not related to metreleptin
Neuropathy peripheral (Nervous system disorders) | 1 — Worsening neuropathy, not related to metreleptin
Anxiety (Psychiatric disorders) | 1 — Worsening of anxiety, not related to metreleptin
Insomnia (Psychiatric disorders) | 1 — Worsening of insomnia, not related to metreleptin
Mental status changes (Psychiatric disorders) | 1 — Altered mental state, not related to metreleptin
Stress (Psychiatric disorders) | 1 — Stress, not related to metreleptin
Acute kidney injury (Renal and urinary disorders) | 1 — Acute kidney injury, not related to metreleptin
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 — FOCAL SEGMENTAL GLOMERULOSCLEROSIS, not related to metreleptin
Bladder spasm (Renal and urinary disorders) | 1 — Bladder spasms, not related to metreleptin
Renal impairment (Renal and urinary disorders) | 1 — DETERIORATING KIDNEY FUNCTION WITH RISING CREATININE, not related to metreleptin
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 — Nose bleed, not related to metreleptin
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 — Sinus congestion, not related to metreleptin
Eczema (Skin and subcutaneous tissue disorders) | 1 — Intermittent scalp eczema, not related to metreleptin
Dermatitis (Skin and subcutaneous tissue disorders) | 1 — Skin rash - dermatitis unspecified
Rash (Skin and subcutaneous tissue disorders) | 1 — Rash on bilateral elbows, not related to metreleptin
Skin lesion (Skin and subcutaneous tissue disorders) | 1 — SKIN LESION EXCISION BY DERMATOLOGY - BENIGN, not related to metreleptin
Urticaria (Skin and subcutaneous tissue disorders) | 1 — Hives, not related to metreleptin
Vitiligo (Skin and subcutaneous tissue disorders) | 1 — Increased vitiligo in mouth, not related to metreleptin
Xanthoma (Skin and subcutaneous tissue disorders) | 1 — Eruptive xanthomas, not related to metreleptin
Abortion induced (Surgical and medical procedures) | 1 — Abortion induced, not related to metreleptin
Arteriovenous fistula (Vascular disorders) | 1 — Arteriovenous fistula, not related to metreleptin

LIMITATIONS AND CAVEATS:
Following limitations may have occurred:

1. Exposure misclassification
2. Selection bias
3. Attrition
4. Confounders (e.g., concomitant use of antidiabetic medications, metreleptin dose and compliance, pregnancy, puberty)
5. Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT04026178/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT04026178/SAP_001.pdf